CLINICAL TRIAL: NCT01317199
Title: Phase I/II Study of Safety and Efficacy of Muscadine Plus (MPX) in Men With Prostate Cancer: a Randomized,Double-blind,Placebo Controlled Study of the Effects of Two Doses of MPX Capsules on Rising Prostate-specific Antigen Levels in Men Following Initial Therapy for Prostate Cancer
Brief Title: Effects of Two Doses of MPX Capsules on Rising Prostate-specific Antigen Levels in Men Following Initial Therapy for Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Howard University (Other); Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J1161
Record Dates: First submitted 2011-03-11; First posted 2011-03-17 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
Keywords: Rising psa
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Arm 1: participants in dose-escalation phase (Phase 1) Arms 2-4: Randomized, double-blind (Phase 2); control, low-dose, high-dose
Who Masked: Participant, Investigator
Masking Description: Phase 1 (Arms 1) - open label Phase 2 (Arms 2-4) - randomized, double-blind
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1: Dose-escalation of Muscadine Plus Grape Skin Extract (Experimental): Muscadine Plus Grape Skin Extract (MPX): Phase I Dose-escalation starts at 500mg daily for 1 cycle (28 days), then increased to 1000mg for 2nd cycle, then increased to 2000mg daily for 3rd cycle, then increased to 3000mg daily for 4th cycle, then increased to maximum dose of 4000mg daily for final cycle. Pills given by mouth once daily for 28 days per cycle.
  Interventions: Drug: Muscadine Plus Grape Skin Extract
- Phase 2: Placebo control (Placebo Comparator): Randomly-assigned participants receive 8 capsules once daily of placebo composed of pulverized rice for up to 12 cycles (28 days per cycle).
  Interventions: Drug: Placebo oral capsule
- Phase 2: Low-dose MPX (Experimental): Randomly-assigned participants receive low-dose (500mg) MPX
  Interventions: Drug: Low-dose MPX
- Phase 2: High-dose MPX (Experimental): Randomly-assigned participants receive high-dose (4000mg) MPX
  Interventions: Drug: High-dose MPX

INTERVENTIONS:
Drug: Muscadine Plus Grape Skin Extract — Phase I: Dose escalation starts at 500mg pills given by mouth once daily for 28 days per cycle
  Arms: Phase 1: Dose-escalation of Muscadine Plus Grape Skin Extract
Drug: Low-dose MPX — Randomly-assigned participants receive one capsule of drug (500mg MPX) and seven capsules of placebo composed of pulverized rice, once daily for up to 12 cycles (28 days per cycle).
  Arms: Phase 2: Low-dose MPX
Drug: High-dose MPX — Randomly-assigned participants receive 8 capsules of drug (4000mg MPX) once daily for up to 12 cycles (28 days per cycle).
  Arms: Phase 2: High-dose MPX
Drug: Placebo oral capsule — Randomly-assigned participants receive 8 capsules once daily of placebo composed of pulverized rice for up to 12 cycles (28 days per cycle).
  Arms: Phase 2: Placebo control

SUMMARY:
This research is being done to test an investigational product called Muscadine Plus in the treatment of men who have received initial therapy (surgery and or radiation, cryotherapy or brachytherapy) for prostate cancer and are experiencing a rise in their prostate-specific antigens (PSA) level.

DETAILED DESCRIPTION:
In phase I the investigators are evaluating the safety of the product and checking blood levels of the active components. In phase II the investigators are evaluating the effect of MPX on PSA doubling time

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Undergone definitive treatment (surgery, surgery with radiation therapy, cryotherapy, radiation therapy or brachytherapy) for the primary prostate tumor.
* Rising PSA on a minimum of 3 time points (including screening psa) within the 12 months prior to study initiation.
* > 18 years of age.
* Life expectancy of greater than 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
* Testosterone level of ≥1.5 ng/mL at screening.
* Adequate kidney, liver and bone marrow function
* Agrees to abstain from other commercially available MP products while participating in this study.
* Subject's use of other dietary/herbal supplements (e.g. saw palmetto, selenium, etc) has been stable for at least 2 months prior to screening and the subject agrees not to stop or change the dose(s) while participating in the study.
* Signed a written informed consent document and agrees to comply with requirements of the study.

Exclusion Criteria:

* Known radiographic evidence of metastatic disease, except for presence of positive lymph nodes from the surgical pathology. Pelvic/intraperitoneal lymph nodes less than 2.0 cm maybe considered nonspecific and the patient would be eligible
* Receipt of any therapies that modulate testosterone levels (e.g., androgen ablative/anti-androgen therapy, 5 alpha reductase inhibitors) for a minimum of 6 months prior to study
* Prior or concomitant treatment with experimental drugs, high dose steroids, or any other cancer treatment within 4 weeks prior to the first dose of the study product
* Consumption of Muscadine Plus over the past 2 months
* Known allergy to muscadine grapes or ellagic acid
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Negative PSA doubling time (1 time point may be excluded per 3e inclusion criteria)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Carducci, MD, Principal Investigator — Johns Hopkins University
Locations (8):
- United States (8):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Howard University College of Medicine, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates:
  Phase I: October 4, 2011-August 7, 2012 in medical clinics Phase II: January 31, 2013-October 20, 2014
Pre-assignment Details: Enrolled subjects agreed to abstain from other commercially available Muscadine Plus products while in this trial.
  If subjects were taking other dietary/herbal supplements (e.g. saw palmetto, selenium, pomegranate juice or pills, etc) prior to study entry, they had to be on a stable dose for 2 months prior and not stop while on trial.
Groups:
- Dose-escalation Phase:Muscadine Plus Grape Skin Extract (MPX): Muscadine Plus Grape Skin Extract: Phase I Dose-escalation starts at 500mg daily for 1 cycle (28 days), then increased to 1000mg for 2nd cycle, then increased to 2000mg daily for 3rd cycle, then increased to 3000mg daily for 4th cycle, then increased to maximum dose of 4000mg daily for final cycle. Pills given by mouth once daily for 28 days per cycle.
- Phase 2: Low-dose MPX: Randomly-assigned participants receive one capsule of drug (500mg MPX) and seven capsules of placebo composed of pulverized rice, once daily for up to 12 cycles (28 days per cycle).
- Phase 2: High-dose MPX: Randomly-assigned participants receive 8 capsules of drug (4000mg MPX) once daily for up to 12 cycles (28 days per cycle).
Period: Dose-escalation Phase 1
Arm/Group | Dose-escalation Phase:Muscadine Plus Grape Skin Extract (MPX) | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Started | 14 | 0 | 0 | 0
Cycle 1: 500mg MPX Once Daily for 28 Day | 2 | 0 | 0 | 0
Cycle 2: 1000mg MPX Daily for 28 Days | 2 | 0 | 0 | 0
Cycle 3: 2000mg MPX Daily for 28 Days | 2 | 0 | 0 | 0
Cycle 4: 3000mg MPX Daily for 28 Days | 2 | 0 | 0 | 0
Cycle 5: 4000mg MPX Daily for 28 Days | 6 | 0 | 0 | 0
Completed | 7 | 0 | 0 | 0
Not Completed | 7 | 0 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0 | 0
Not completed — Disease progression | 1 | 0 | 0 | 0
Not completed — Comorbidities, myasthenia gravis | 1 | 0 | 0 | 0
Period: Randomized Phase 2
Arm/Group | Dose-escalation Phase:Muscadine Plus Grape Skin Extract (MPX) | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Started | 0 | 24 | 56 | 49
Completed | 0 | 13 | 35 | 32
Not Completed | 0 | 11 | 21 | 17
Not completed — Disease progression | 0 | 3 | 7 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Comorbidities | 0 | 2 | 2 | 2
Not completed — Rising PSA, not as defined by protocol | 0 | 2 | 5 | 2
Not completed — Disenrolled before treatment | 0 | 1 | 1 | 2
Not completed — Patient stopped taking study drug | 0 | 0 | 0 | 1
Not completed — Patient transferred to other facility | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Phase:Muscadine Plus Grape Skin Extract (MPX) | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX | Total
Number analyzed (Participants) | 14 | 24 | 56 | 49 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (7.5) | 69 (7.1) | 67 (7.2) | 68 (6.9) | 67.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 14 | 24 | 56 | 49 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 12 | 10 | 32
  White | 10 | 18 | 43 | 38 | 109
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 24 | 56 | 49 | 143
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) scale is a measure of performance status with 0 (fully active) as the best score and 1 being restricted to physically strenuous activity. Population: Baseline characteristics were not collected for subjects who withdrew from the study. ECOG was not analyzed in the dose-escalation phase.
  Participants
    number analyzed (Participants) | 0 | 23 | 54 | 47 | 124
    0 |  | 18 | 52 | 39 | 109
    1 |  | 5 | 2 | 8 | 15
Gleason score [Count of Participants; unit: Participants] — The gleason score is an indication of prognosis based on prostate pathology. The score ranges from 2 to 10 with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5). Population: Gleason score was recorded differently in the dose-escalation phase and phase 2.
  Participants
    ≤6, 3+4: number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    ≤6, 3+4 |  | 11 | 25 | 23 | 59
    ≥8, 4+3: number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    ≥8, 4+3 |  | 13 | 31 | 26 | 70
    6: number analyzed (Participants) | 14 | 0 | 0 | 0 | 14
    6 | 3 |  |  |  | 3
    7: number analyzed (Participants) | 14 | 0 | 0 | 0 | 14
    7 | 7 |  |  |  | 7
    8: number analyzed (Participants) | 14 | 0 | 0 | 0 | 14
    8 | 1 |  |  |  | 1
    9: number analyzed (Participants) | 14 | 0 | 0 | 0 | 14
    9 | 3 |  |  |  | 3
Baseline PSA doubling time (PSADT) [Mean (Standard Deviation); unit: months] — Population: Baseline PSADT was recorded as a mean in the dose-escalation phase, versus as number of participants with greater than or less than 9 months PSADT in Phase 2.
  months
    number analyzed (Participants) | 14 | 0 | 0 | 0 | 14
    (all) | 13 (10.1) |  |  |  | 13 (10.1)
Baseline PSADT [Count of Participants; unit: Participants] — Population: Baseline PSADT was recorded as a mean in the dose-escalation phase, versus as number of participants with greater than or less than 9 months PSADT in Phase 2.
  Participants
    number analyzed (Participants) | 0 | 23 | 55 | 48 | 126
    ≤9 months |  | 13 | 32 | 27 | 72
    >9 months |  | 10 | 23 | 21 | 54
Prior therapy [Count of Participants; unit: Participants] — Population: Participants in Phase 2 were not categorized as 'Radiation & Surgery'. Only individual counts for each prior therapy received was recorded.
  Participants
    Radiation | 4 | 21 | 49 | 42 | 116
    Surgery | 1 | 16 | 40 | 32 | 89
    Radiation & Surgery: number analyzed (Participants) | 14 | 0 | 0 | 0 | 14
    Radiation & Surgery | 9 |  |  |  | 9
    Cryotherapy: number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    Cryotherapy |  | 0 | 49 | 1 | 50
    Brachytherapy: number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    Brachytherapy |  | 3 | 5 | 3 | 11
    Androgen Deprivation Therapy (ADT): number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    Androgen Deprivation Therapy (ADT) |  | 2 | 25 | 19 | 46
Superoxide dismutase 2 (SOD2) genotype [Count of Participants; unit: Participants] — Population: SOD2 genotype was not recorded in dose-escalation phase. In Phase 2, SOD2 genotype was not recorded for all participants if data was unavailable.
  Participants
    Alanine/Alanine (Ala/Ala): number analyzed (Participants) | 0 | 21 | 44 | 37 | 102
    Alanine/Alanine (Ala/Ala) |  | 5 | 12 | 10 | 27
    Alanine/Valine (Ala/Val): number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    Alanine/Valine (Ala/Val) |  | 11 | 21 | 22 | 54
    Valine/Valine (Val/Val): number analyzed (Participants) | 0 | 24 | 56 | 49 | 129
    Valine/Valine (Val/Val) |  | 5 | 11 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: (Phase I) Maximum Tolerated Dose
Description: To determine the recommended dosing for Muscadine Plus and to evaluate the safety and tolerability of Muscadine Plus in prostate cancer patients with rising PSA following definitive therapy.
Time Frame: Up to 7 months post-intervention
Measure: Number; unit: mg
Arm/Group | Dose-escalation Phase:Muscadine Plus Grape Skin Extract (MPX) | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Number analyzed (Participants) | 14 | 0 | 0 | 0
mg | 4000 |  |  |

2. Primary Outcome: (Phase II) Prostate Specific Antigen Doubling Time (PSADT)
Description: To define the effects of placebo and two different daily doses of MPX on PSADT in men who have rising PSA after initial definitive therapy for localized prostate cancer.
Time Frame: Change from baseline to month 12
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Number analyzed (Participants) | 20 | 52 | 40
months | 0.9 [-6.7 to 83.1] | 1.5 [-10.3 to 87.2] | 0.9 [-27.3 to 88.1]

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events reported verbally by patient and documented in study notes.
Time Frame: At month 12 post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Phase:Muscadine Plus Grape Skin Extract (MPX) | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Number analyzed (Participants) | 14 | 23 | 55 | 47
Participants | 7 | 19 | 38 | 32

4. Secondary Outcome: (Phase II) Proportion of Men Whose PSADT Increases Greater Than 33%
Time Frame: At month 12 post-intervention
Population: Data was not collected for this secondary outcome measure.
Arm/Group | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: (Phase II) Number of Men With Greater Than 50% Reduction in PSA Compared to Baseline
Description: Change in PSA values drawn over study period, taken every 3 months. PSA is measured in ng/mL
Time Frame: At month 12 post-intervention
Population: Patients counted in the analysis were evaluable if they completed at least six cycles of treatment prior to discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
Number analyzed (Participants) | 20 | 52 | 40
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Groups:
- Phase 1:Muscadine Plus Grape Skin Extract (MPX) 500mg; Dose-escalation Phase 1: MPX 1000mg; Dose-escalation Phase 1: MPX 2000mg; Dose-escalation Phase 1: MPX 3000mg; Dose-escalation Phase 1: MPX 4000mg: Muscadine Plus Grape Skin Extract: Phase I Dose-escalation starts at 500mg daily for 1 cycle (28 days), then increased to 1000mg for 2nd cycle, then increased to 2000mg daily for 3rd cycle, then increased to 3000mg daily for 4th cycle, then increased to maximum dose of 4000mg daily for final cycle. Pills given by mouth once daily for 28 days per cycle.
Arm/Group | Phase 1:Muscadine Plus Grape Skin Extract (MPX) 500mg | Dose-escalation Phase 1: MPX 1000mg | Dose-escalation Phase 1: MPX 2000mg | Dose-escalation Phase 1: MPX 3000mg | Dose-escalation Phase 1: MPX 4000mg | Phase 2: Placebo Control | Phase 2: Low-dose MPX | Phase 2: High-dose MPX
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/6 | 0/23 | 0/55 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/6 | 0/23 | 1/55 | 1/47
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/2 | 0/2 | 3/6 | 3/23 | 10/55 | 7/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1:Muscadine Plus Grape Skin Extract (MPX) 500mg (N=2) | Dose-escalation Phase 1: MPX 1000mg (N=2) | Dose-escalation Phase 1: MPX 2000mg (N=2) | Dose-escalation Phase 1: MPX 3000mg (N=2) | Dose-escalation Phase 1: MPX 4000mg (N=6) | Phase 2: Placebo Control (N=23) | Phase 2: Low-dose MPX (N=55) | Phase 2: High-dose MPX (N=47)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug.
Vocal Chord Squamous Cell Carcinoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1:Muscadine Plus Grape Skin Extract (MPX) 500mg (N=2) | Dose-escalation Phase 1: MPX 1000mg (N=2) | Dose-escalation Phase 1: MPX 2000mg (N=2) | Dose-escalation Phase 1: MPX 3000mg (N=2) | Dose-escalation Phase 1: MPX 4000mg (N=6) | Phase 2: Placebo Control (N=23) | Phase 2: Low-dose MPX (N=55) | Phase 2: High-dose MPX (N=47)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 6 (6) | 3 (3) — Related to study drug
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes